CLINICAL TRIAL: NCT05017753
Title: Thoracentesis to Alleviate Cardiac Pleural Effusion - an Interventional Trial (TAP-IT)
Brief Title: Thoracentesis to Alleviate Cardiac Pleural Effusion
Acronym: TAP-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Independent Research Fund Denmark (Industry); Hartmann Fonden (Other); University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Jens Jakob Thune, Clinical Research Associate Professor, Consultant Cardiologist, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAP-IT
Record Dates: First submitted 2021-08-12; First posted 2021-08-24 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure; Pleural Effusion
Keywords: Heart failure; Systolic heart failure; Pleural effusion; Thoracentesis; Thoracocentesis; Pleurocentesis
MeSH Terms: conditions — Heart Failure; Pleural Effusion; Heart Failure, Systolic | interventions — Thoracentesis

STUDY DESIGN:
Intervention Model Description: The trial is a pragmatic controlled, randomized, multicenter open label trial with including patients admitted with pleural effusion related to systolic heart failure. Patients will be randomized 1:1 to standard-of-care medical treatment only or standard-of-care medical treatment and referral to thoracentesis. Randomization will be stratified according to whether patients are treated with oral anticoagulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Standard-of-care medical treatment.
  Interventions: Drug: Standard-of-care medical treatment
- Intervention group (Experimental): Thoracentesis in addition to standard-of-care medical treatment.
  Interventions: Procedure: Thoracentesis

INTERVENTIONS:
Procedure: Thoracentesis — Thoracentesis will be performed according to local practice, either at the ward or at the radiology department, in addition to standard-of-care medical treatment.
  Other Names: Thoracocentesis; Pleurocentesis
  Arms: Intervention group
Drug: Standard-of-care medical treatment — Standard-of-care medical treatment
  Arms: Control group

SUMMARY:
The present study will examine the comparative effectiveness of two treatment strategies currently used in the treatment of patients with systolic heart failure presenting with pleural effusion. Patients will be randomized to standard medical treatment only or medical treatment and referral to thoracentesis.

Study hypothesis: A strategy of referring patients with heart failure-related pleural effusion to thoracentesis increases number of days alive outside of hospital over the following 90 days.

DETAILED DESCRIPTION:
Purpose and Rationale: Pleural effusion is a common presentation in patients with heart failure, and the condition is related to a poor prognosis and increased mortality. Therapeutic options consist of intensification of diuretic treatment and invasive drainage of the effusion (thoracentesis). Thoracentesis is a common medical procedure and is often performed on patients with heart failure presenting with a pleural effusion, but there is no randomized evidence to guide the use of thoracentesis in heart failure-related pleural effusion. International guidelines provide no recommendations. Some Danish hospitals use thoracentesis frequently, some rarely. Hence, there is true clinical equipoise and a strong need to assess whether thoracentesis benefits patients or not.

Study Hypothesis: A strategy of referring patients with heart failure-related pleural effusion to thoracentesis increases number of days alive outside of hospital over the following 90 days.

Study Setting:126 adult patients admitted with systolic heart failure and pleural effusion documented by either chest x- ray, ultrasound, computed tomography (CT) or magnetic resonance imaging (MRI) will be randomized 1:1 to medical treatment only or medical treatment and referral to thoracentesis. Thoracentesis will be performed according to local practice. Randomization will be stratified according to whether patients are treated with oral anticoagulation.

Crossover/rescue thoracentesis: For patients in the medical treatment arm whose condition deteriorates to the degree that the participant fulfill any of the study exclusion criteria (eg. increased need of oxygen), thoracentesis may be performed immediately. Some patients randomized to medical treatment only may prove to be too diuretic resistant to achieve an adequate effect of medical treatment alone. The recommended waiting period before performing thoracentesis on a patient in the control group is 5 days from randomization.

Patients may be discharged at the discretion of the treating physician. The follow up period is planned to 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction (LVEF) ≤ 45%
* Non- negligible pleural effusion by x-ray, ultrasound, CT or MRI, suspected to be due to heart failure
* Age ≥ 18 years

Exclusion Criteria:

* Clinically indicated diagnostic thoracentesis (e.g. suspected malignant aetiology)
* Suspected pulmonary or pleural infection (pneumonia symptoms with c- reactive protein>100 mg/L or white blood count>11)
* Recent (<3 months) intrathoracic procedure (including heart or lung surgery, transcatheter aortic valve implantation (TAVI) or thoracentesis)
* Contraindications to thoracentesis according to local guidelines (such as spontaneously elevated international normalized ratio (INR) or thrombocytopenia), patients on oral anticoagulation may be randomized.
* Severe aortic stenosis
* Massive pleural effusion (equivalent to >2/3 of lung on a standing chest x-ray)
* Substantially affected hemodynamics (systolic blood pressure < 85mmHg, need of inotropes) or high oxygen demand (>7L/min)
* Estimated glomerular filtration rate (eGFR) <15ml/min/1.73m2 or dialysis treatment
* Planned or expected admission > 10 days for other condition than heart failure
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Days alive outside of hospital (days) | 90 days
  Number of days the patient is alive outside of hospital in the 90 days following randomization

SECONDARY OUTCOMES:
Satisfaction with hospital stay (Likert scale) | Up til 1 week after discharge
  Selected questions from the questionnaire "Questions about your admission" from the annual Danish National Survey of Patient Experiences to assess satisfaction with index admission. Likert scale from 1-5. 5 represents the best outcome.
Kansas City Cardiomyopathy Questionnaire (KCCQ-23) (score) | At 14 days and 90 days - up til 1 week
  Kansas City Cardiomyopathy Questionnaire (KCCQ). Selected scores from the 23-item questionnaire at 14 and 90 days. Scores from 0-100 with 100 representing the best outcome.
Complications during hospital stay (count) | From randomization until the date af discharge from hospital. Estimated time frame from 2 days to 3 weeks.
  Number of complications during the index admission (eg. infections, delirium, falls, thrombosis)
Complications to thoracentesis (count) | From randomization until the date af discharge from hospital. Estimated time frame from 2 days to 3 weeks.
  Number of complications to interventional thoracentesis
Duration of index admission (days) | From randomization until the date af discharge from hospital. Estimated time frame from 2 days to 3 weeks.
  Duration of index admission following randomization.
Changes from baseline in weight during admission (kg) | From randomization until the date af discharge from hospital. Estimated time frame from 2 days to 3 weeks.
  Changes in weight during admission
Change from baseline in dosage of diuretics during admission (mg/day) | From randomization until the date af discharge from hospital. Estimated time frame from 2 days to 3 weeks.
  Change in dosage of diuretics during index admission
Time to death (days) | 90 days
Time to first readmission or death (days) | 90 days
Days alive and not hospitalized due to heart failure during the 90 days following randomization. | 90 days

CONTACTS AND LOCATIONS:
Locations (10):
- Denmark (10):
  - University Hospital Aalborg, Aalborg
  - University Hospital Aarhus, Aarhus
  - University Hospital Bispebjerg and Frederiksberg, Copenhagen
  - University Hospital Rigshospitalet, Copenhagen
  - University Hospital Rigshospitalet, Glostrup, Glostrup Municipality
  - University Hospital Herlev/Gentofte, Herlev
  - University Hospital Nordsjaelland, Hillerød
  - University Hospital Hvidovre, Hvidovre
  - University Hospital Odense, Odense
  - University Hospital Zealand, Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: Yes
De-identified data necessary to reproduce published results will be made available on reasonable requests.

REFERENCES:
- [Derived] Glargaard S, Thomsen JH, Tuxen C, Lindholm MG, Bang CA, Schou M, Iversen K, Rasmussen RV, Logstrup BB, Vraa S, Stride N, Seven E, Barasa A, Tofterup M, Hofsten DE, Rossing K, Kober L, Gustafsson F, Thune JJ. A Randomized Controlled Trial of Thoracentesis in Acute Heart Failure. Circulation. 2025 Apr 22;151(16):1150-1161. doi: 10.1161/CIRCULATIONAHA.124.073521. Epub 2025 Apr 1. PMID 40166829
- [Derived] Glargaard S, Thomsen JH, Logstrup BB, Schou M, Iversen KK, Tuxen C, Nielsen OW, Bang CA, Lindholm MG, Seven E, Barasa A, Stride N, Vraa S, Tofterup M, Rasmussen RV, Hofsten DE, Rossing K, Kober L, Gustafsson F, Thune JJ. Thoracentesis to alleviate pleural effusion in acute heart failure: study protocol for the multicentre, open-label, randomised controlled TAP-IT trial. BMJ Open. 2024 Jan 19;14(1):e078155. doi: 10.1136/bmjopen-2023-078155. PMID 38245015

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT05017753/SAP_001.pdf